CLINICAL TRIAL: NCT03990987
Title: The Effect of Intraoperative Use of Dexmedetomidine During the Daytime Operation vs the Nighttime Operation on Postoperative Sleep Quality and Pain Under General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Other Study IDs: Dexmedetomidine and sleep
Record Dates: First submitted 2019-06-11; First posted 2019-06-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain; Postoperative Sleep Quality; Intraoperative Dexmedetomidine; General Anesthesia
Keywords: postoperative pain; postoperative sleep quality; dexmedetomidine; general anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Day group: patients in Day group accept operation from 8：00～12：00
  Interventions: Other: time of receiving operation
- Night group: patients in Night group accept operation from 18：00～22：00
  Interventions: Other: time of receiving operation

INTERVENTIONS:
Other: time of receiving operation — patients were randomly divided into Day group (D group) (8：00～12：00) and Night group (N group) (18：00～22：00), Patients received propofol, remifentanil, and DEX for general anesthesia maintenance

SUMMARY:
General anesthesia is a medically induced state of low reactivity consciousness which is similar to natural sleep. Some studies found that general anesthesia as an independent risk factor could result in a desynchronization of the circadian time structure and cause postoperative sleep disorders characterized by reduced rapid eye movement (REM) and slow wave sleep (SWS), which have signiﬁcant deleterious impacts on postoperative outcomes, such as postoperative fatigue, severe anxiety and depression, emotional detachment and delirium, and even pain sensitivity or postoperative pain of patients.Clinical trials have already proved that intraoperative use of dexmedetomidine (DEX) for general anesthesia, a highly selective alpha-2 adrenergic agonist, was able to improve sedative and analgesia effects and promote sleep quality (by decreasing stage N1 sleep, increasing stage N2 sleep and sleep efficiency). However, Wenfei Tan et al reported that with the deeper sedative state provided by DEX in the daytime, the elderly male patients undergoing TURP under spinal anesthesia suffered worse sleep on the night of surgery. Thus, what the effect of intraoperative using DEX at different time periods under general anesthesia on postoperative sleep quality and pain will be needs further study.

DETAILED DESCRIPTION:
patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were enrolled. Patients were randomized to receive operation in the D group (8:00-12:00) and the N group (18:00-22:00). The Portable Sleep Monitor (PSM) was performed on the following 3 nights: the night before surgery (Sleep1), the ﬁrst night after surgery (Sleep 2), and the third night after surgery (Sleep 3). Postoperative pain scores using visual analogue scoring scale, subjective sleep quality using the Athens Insomnia Scale, total dose of general anesthetics and PCA pump press numbers were also recorded.

ELIGIBILITY:
Inclusion Criteria:

age between 30 and 55 years American Society of Anaesthesiologists physical status I or II.

Exclusion Criteria:

cardiovascular disease long term use of analgesia preoperative heart rate (HR) less than 50 beats/min second- or third-degree atrioventricular block sleep disorder sleep apnea syndrome history of abnormal operation or anesthesia recovery psychosis or a patient with a language communication disorder not willing to cooperate with the experimenter.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who underwent elective laparoscopic abdominal surgeries under general anesthesia at Shengjing Hospital of China Medical University were enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep quality of one night before the surgery | one night before the surgery
  Use sleep monitor to test the sleep quality on one night before the surgery
Sleep quality of first night after the surgery | the first night after the surgery
  Use sleep monitor to test the sleep quality on the first night after the surgery
Sleep quality of third night after the surgery | the third night after the surgery
  Use sleep monitor to test the sleep quality on the third night after the surgery

SECONDARY OUTCOMES:
Visual analog scale (VAS) | 1,6,24,48 hours after the surgery
  Evaluate the VAS score at 1,6,24,48 hours after the surgery.Visual analog scale (VAS) score of 0 was considered painless, and a score of 10 was considered as intense pain. Scores of 4 and below were considered mild pain (pain does not affect sleep), and scores of 5 to 6 were considered moderate pain (pain influences sleep, but the patients can still fall asleep). Scores of 7 and above were considered severe pain (Due to the pain the patient is unable to sleep or wakes up)
PCA pump press number | 48 hours after the surgery
  Evaluate the Pump press number 48 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, Study Director — Shengjing Hospital
Locations (1):
- shengjing hospital of China medical university, Shenyang, Liaoning, China